CLINICAL TRIAL: NCT01720043
Title: Hemostatic Effects of VELCADE®* Treatment in Multiple Myeloma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI57748
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All participants (Experimental): All participants enrolled
  Interventions: Drug: Velcade

INTERVENTIONS:
Drug: Velcade — Single dose of Velcade (1.0-1.3 mg/m2 dose)
  Other Names: Bortezomib

SUMMARY:
To evaluate the effect of VELCADE on platelet aggregation at baseline, 24 hours and 48 hours after infusion in patients with multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of multiple myeloma
* Patients should have not have received VELCADE for at least 2 weeks before receiving treatment with VELCADE for platelet aggregation testing
* Patients are to be instructed not to take aspirin or ibuprofen 7-10 days prior to the platelet aggregations testing.
* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice 2 effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of VELCADE, or agree to completely abstain from heterosexual intercourse.
* Male subjects, even if surgically sterilized (ie, status postvasectomy) must agree to 1 of the following: practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, or completely abstain from heterosexual intercourse.

Exclusion Criteria:

* Patients who have received Velcade within 2 weeks prior to study registration
* Patient has a platelet count of < 150,000 within 7 days before enrollment.
* Patient has an absolute neutrophil count of < 1000 within 7 days before enrollment.
* Patient has > 1.5 x ULN Total Bilirubin
* Patient has > Grade 2 peripheral neuropathy
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* Currently receiving medication with Coumadin, heparin, low molecular weight heparin, or NSAIDS. Concomitant use with any of these medications must be discontinued within two weeks prior to beginning protocol treatment.
* Patient has hypersensitivity to VELCADE, boron, or mannitol.
* Female subject is pregnant or lactating. Confirmation that the subject is not pregnant must be established by a negative serum pregnancy test result obtained during screening. Pregnancy testing is not required for postmenopausal or surgically sterilized women.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on Day 1 before first dose of study drug, if applicable.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tibor Kovacsovics, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Velcade
Description: Effect of VELCADE at 1.0-1.3 mg/m2 dose on platelet aggregation at 24 and 48 hour post-infusion in patients with multiple myeloma. The following components of platelet aggregation were evaluated at varying levels: Collagen, Adenine di-Phosphate (ADP), Arachidonic acid, and Ristocetin.
Time Frame: 48 hours
Population: One patient withdrew before receiving the 24 hour dose, leaving 7 patients evaluable for response.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | All Participants
Number analyzed (Participants) | 7
percentage
  Collagen 5.g.ml, 24 hrs | -4.143 (7.244)
  Collagen 2.g.ml, 24 hrs | -4.429 (7.390)
  ADP.10.M, 24 hrs | -4.571 (6.949)
  ADP.5.M, 24 hrs | -6.429 (7.591)
  ADP.3.M, 24 hrs | -7.571 (16.400)
  Arach.Acid.0.5.mg.ml, 24 hrs | -11.143 (15.507)
  Ristocetin1.5.mg.ml, 24 hrs | -1.429 (7.345)
  Ristocetin.0.5.mg.ml, 24 hrs | -2.429 (6.803)
  Collagen.5.g.mL, 48 hrs | -2.429 (10.130)
  Collagen.2.g.mL, 48 hrs | -0.857 (10.605)
  ADP.10.M, 48 hrs | -3.429 (7.044)
  ADP.5.M, 48 hrs | -3.571 (10.845)
  ADP.3.M, 48 hrs | 1.571 (13.587)
  Arach.Acid.0.5.mg.mL, 48 hrs | -2.286 (11.368)
  Ristocetin.1.5.mg.mL, 48 hrs | .0143 (9.353)
  Ristocetin.0.5.mg.mL, 48 hrs | -2.000 (4.041)
Statistical Analysis 1: Comparison: All Participants; Collagen.5.g.ml, 24 hrs; Test type: Superiority; p = 0.181, t-test, 2 sided
Statistical Analysis 2: Comparison: All Participants; Collagen.2.g.ml; Test type: Superiority; p = .164, t-test, 2 sided
Statistical Analysis 3: Comparison: All Participants; ADP.10.M, 24 hrs; Test type: Superiority; p = .132, t-test, 2 sided
Statistical Analysis 4: Comparison: All Participants; ADP.5.M; Test type: Superiority; p = .066, t-test, 2 sided
Statistical Analysis 5: Comparison: All Participants; ADP.3.M, 24 hrs; Test type: Superiority; p = 0.268, t-test, 2 sided
Statistical Analysis 6: Comparison: All Participants; Arach.Acid.0.5.mg.ml; Test type: Superiority; p = 0.106, t-test, 2 sided
Statistical Analysis 7: Comparison: All Participants; Ristocetin.1.5.mg.ml; Test type: Superiority; p = 0.625, t-test, 2 sided
Statistical Analysis 8: Comparison: All Participants; Ristocetin.0.5.mg.ml; Test type: Superiority; p = 0.381, t-test, 2 sided
Statistical Analysis 9: Comparison: All Participants; Collagen.5.g.ml, 48 hrs; Test type: Superiority; p = 0.549, t-test, 2 sided
Statistical Analysis 10: Comparison: All Participants; Collagen.2.g.ml, 48 hrs; Test type: Superiority; p = .838, t-test, 2 sided
Statistical Analysis 11: Comparison: All Participants; ADP.10.M; Test type: Superiority; p = 0.245, t-test, 2 sided
Statistical Analysis 12: Comparison: All Participants; ADP.5.M; Test type: Superiority; p = 0.417, t-test, 2 sided
Statistical Analysis 13: Comparison: All Participants; ADP.3.M, 48 hrs; Test type: Superiority; p = 0.770, t-test, 2 sided
Statistical Analysis 14: Comparison: All Participants; Arach.Acid.0.5.mg.ml, 48 hrs; Test type: Superiority; p = 0.614, t-test, 2 sided
Statistical Analysis 15: Comparison: All Participants; Ristochetin.1.5.mg.ml; Test type: Superiority; p = 0.969, t-test, 2 sided
Statistical Analysis 16: Comparison: All Participants; Ristocetin.0.5.mg.ml, 48 hrs; Test type: Superiority; p = 0.238, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=8)
Pain (General disorders) | 1 (1)
DVT (Vascular disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No